CLINICAL TRIAL: NCT05730595
Title: A Randomized Controlled Trial of Fluorescence Laparoscopic Navigation of the Extent of Lymph Node Dissection for High Rectal Cancer and Sigmoid Colon Cancer
Brief Title: Fluorescence Laparoscopic Navigation for Rectal Cancer and Sigmoid Colon Cancer
Acronym: FLORA-01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Fudan University (Other); Fujian Province Tumor Hospital (Other); Guangdong Provincial People's Hospital (Other); Shengjing Hospital (Other); Affiliated Hospital of Qinghai University (Other); Hebei Medical University Fourth Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Jiangxi Provincial Cancer Hospital (Other); The First Hospital of Jilin University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Shanxi Province Cancer Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Second People's Hospital of Yunnan Province (Other); Binzhou Medical University (Other); The First Affiliated Hospital of University of Science and Technology of China (Other); First Affiliated Hospital of Chengdu Medical College (Other); The Second People's Hospital of Yibin (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jianqiang Tang, Associate professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCC20231
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Neoplasms; Fluorescence; Lymph Node Excision
Keywords: Colorectal cancer; Fluorescence laparoscopic navigation; Lymph node dissection
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lymph Node Excision

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D2 lymph node dissection (Experimental): The D2 lymph node region are dissected. And 1-3 lymph nodes of the D2 region will be selected for intraoperative frozen section. If no lymph node metastasis is found in freezing, the D3 region lymph nodes in the root of the submesenteric artery were preserved.
  Interventions: Procedure: lymph node dissection
- D3 lymph node dissection (Active Comparator): Thorough dissection of lymph nodes in the D3 region.
  Interventions: Procedure: lymph node dissection

INTERVENTIONS:
Procedure: lymph node dissection — The extent of lymph node dissection varies between groups
  Other Names: Fluorescence-guided laparoscopic surgery; Radical operation for rectal cancer and sigmoid Cancer

SUMMARY:
To explore the short-term and long-term outcomes of fluorescence laparoscopic navigation D2 lymph node dissection for colorectal cancer surgery by comparing it with D3 lymph node dissection.

DETAILED DESCRIPTION:
Lymph node metastasis is the most common metastatic mechanisms for colorectal cancer. Therefore, regional lymph node dissection is the key part in radical surgery for colorectal cancer. In patients who have developed lymph node metastases, inadequate lymph node dissection will promote tumor recurrence. In patients who do not develop lymph node metastases, excessive lymph node dissection not only does not improve the patient's prognosis, but also increases surgical trauma and destroys the antitumor effect of the lymphoid immune system. There is still some controversy over whether to choose D3 lymph node dissection or D2 lymph node dissection for rectal and sigmoid cancer. Fluorescence laparoscopic navigation techniques can guide lymph node dissection by visualizing lymph nodes more clearly during surgery.

This study will compare the short-term and long-term oncological outcomes between fluorescence laparoscopic navigation D2 and D3 lymph node dissection by conducting a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants are aged 18-75;
* Colonoscopy biopsy confirms colorectal adenocarcinoma;
* Colonoscopy shows that the lower edge of the tumor is located more than 10 cm from the margin or the tumor is located in the upper rectum and sigmoid colon by imaging diagnosis;
* The tumor is staged cT1-4aNxM0 by preoperative imaging;
* Participants have no local complications before surgery.

Exclusion Criteria:

* Previous history of malignant colorectal tumor;
* Multiple primary colorectal tumors;
* Preoperative imaging reveals suspicious positive lymph nodes in the submesenteric artery root region (area 253);
* Patients undergoing neoadjuvant therapy before surgery;
* With contraindications to laparoscopic surgery;
* Histoty of multiple abdominal and pelvic surgery or extensive abdominal adhesions;
* Other malignancies were diagnosed within the past 5 years;
* History of severe mental illness;
* Pregnant or lactating women;
* With uncontrolled infection before surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | The endpoint of the disease-free survival assessment is the last follow-up or disease recurrence. Follow-up time is up to 36 months.
  Disease-free survival is defined as the time from the surgery to disease recurrence or last follow-up, which was measured in months.
Overall survival | The endpoint of the overall survival assessment is the last follow-up or patient death. Follow-up time is up to 36 months.
  Overall survival is defined as the time from the surgery to death or last follow-up, regardless of disease recurrence, which was measured in months.

SECONDARY OUTCOMES:
The number of lymph node resection | Until the pathological result is available , an average of 14 days.
  The number of lymph nodes removed during surgery, which is obtained by postoperative pathological results
Blood loss | Until the end of the operation, an average of 8 hours.
  Blood loss is defined as intraoperative blood loss and measured in milliliters(ml).
Complications | Until the patient recovered and was discharged from the hospital, an average of 10 days.
  Complications are defined as all surgery-related adverse events postoperatively, such as anastomotic leak, infection, which are measured in frequency.
Hospital stay after surgery | Until the patient recovered and was discharged from the hospital, an average of 10 days.
  Hospital stay after surgery is defined as the length of time from the end of surgery
Function score | Until one year after the patient's surgery
  Function score includes International Prostate Symptom Score, low anterior resection syndrome score and International Index of Erectile Function-5 score, which are used for assess the physical function.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Chengdu
  - Fujian Province Tumor Hospital, Fuzhou, Fujian
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangxi Provincial Cancer Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital, Shenyang, Liaoning
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Binzhou Medical University, Binzhou, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - The second People's Hospital of Yunnan Province, Kunming, Yunnan